CLINICAL TRIAL: NCT02541175
Title: Paroxysmal Atrial Fibrillation Detection and Heart Beat Classification in Multi-Channel Esophageal Long-Term ECG
Brief Title: Multi-Channel Esophageal ECG Signal Classification
Acronym: MC-EECG
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Bern University of Applied Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 149/15
Record Dates: First submitted 2015-08-27; First posted 2015-09-04 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Atrial Fibrillation; Atrial Function; Arrhythmias, Cardiac; Atrial Premature Complexes
Keywords: Electrocardiography; Automation; Arrhythmias, Cardiac; Atrial Fibrillation; Atrial Flutter; Atrial Premature Complexes; Esophagus
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Atrial Premature Complexes; Atrial Flutter

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All study participants: In order to cover a wide variety of common arrhythmias but keeping the number of subjects needed low (pilot study), the subjects are pre-selected according to following 4 categories: 1) 4 patients with intermitting or persisting atrial fibrillation. 2) 4 patients with atrial flutter 3) 6 patients with frequent atrial or ventricular extra-systoles. 4) 6 cardiac healthy subjects.

SUMMARY:
This study is designed to prove new methods to enable the automated analysis of esophageal electrocardiography (eECG) signals in long-term measurements as well as the detection of atrial fibrillation. The investigators hypothesis is that eECG signals allow the reliable atrial and ventricular ECG signal distinction and the detection of atrial fibrillation. Therefore 14 patients with arrhythmias and 6 cardiac healthy subjects are asked to take part in this study. On each subject an esophageal ECG and a simultaneous standard surface ECG will be taken for about half an hour. Patient undergoing a cardiac catheter ablation during their current hospitalization will be further asked to allow access to the invasively obtained measurements (i.e. atrial potential map) to further improve the understanding of the eECG signals.

DETAILED DESCRIPTION:
Background

The fast and correct diagnosis of heart rhythm disorders is very important to reduce morbidity and mortality in cardiovascular patients. Atrial fibrillation is of special interest, because it is an important cause of devastating brain strokes. A significant number of strokes have a cardioembolic genesis due to paroxysmal atrial fibrillation which was not diagnosed early enough. Therefore, it is very important to detect atrial fibrillation as soon as possible. With oral anticoagulation an effective therapeutic option in available to prevent cardioembolisms.

In the clinical routine, mostly 24-hour or 7-day ECGs are made to look for cardiac arrhythmias. The use of such devices is well established. Nevertheless, they have some side effects/limitations. Skin electrodes used for derivation of the ECG often cause skin irritation, sometimes leading to premature termination of the recording. Because of dryout of the contact gel (causes artifacts), small p-waves and especially also motion artifacts, triggered recording or semi-automatic analysis of the recording is problematic, but for longer recording times such a semi-automatic analysis would be helpful. As an alternative esophageal electrocardiography can be performed. Signal quality of the ECG recording (especially of the left atrium) is better than in the standard surface ECG because of the vicinity of the esophagus and the left atrium. The esophagus tolerates well foreign bodies as the investigators know from long-term nasogastric intubation. Therefore use of the esophageal technique for long-term rhythm monitoring is an interesting and promising alternative to conventional surface Holter ECGs.

Earlier studies have already shown the improved p-wave in eECG signals, but the automatic or semi-automatic wave analysis algorithms were not satisfactory. By increasing the number of measuring channels on the esophageal catheter, new classes of algorithm can be applied in order to increase the detection reliability. Using multiple channels to increase the quality of the result is an intuitive and widely used method e.g. in 12 lead ECG or EECG, etc.

Objective

Primary Objective: Differentiation of electrical atrial and ventricular cardiac activity (A/V classification) Secondary Objective: Detection of atrial fibrillation sequences (AFib Detection)

Methods

20 subjects are included in this pilot study to verify enhanced multi-channel detection algorithm. In order to cover a wide variety of arrhythmias to test the algorithm with, the subjects are selected according to 4 categories: 1) 4 patients with intermitting or persisting atrial fibrillation. 2) 4 patients with atrial flutter 3) 6 patients with frequent atrial or ventricular extra-systoles. 4) 6 cardiac healthy subjects. In total around 50'000 heart beats are recorded. The surface ECG signal is used as the reference (manually analyzed). Sensitivity and specificity of the correctly detected atrial and ventricular activities compared to this manual reference including the 95% confidence intervals are calculated (A/V Classification). Additionally the sensitivity and specificity of the detected of atrial fibrillation sequences including the 95% confidence intervals are calculated (AFib Detection).

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years
* Written informed consent
* ambulatory/hospitalized due to peripheral percutaneous intervention
* ambulatory/hospitalized due to shunt stenosis or occlusion
* ambulatory/hospitalized due to electrophysiological intervention
* ambulatory/hospitalized due to pacemaker implantation
* ambulatory/hospitalized due to decompensated heart failure
* ambulatory/hospitalized due to planed cardioangiography
* ambulatory/hospitalized due to performed cardioangiography after Non-ST-elevation myocardial infarction (NSTEMI) or ST-elevation myocardial infarction (STEMI)
* cardiac healthy adults

Exclusion Criteria

* History of ablation of atrial fibrillation
* History of heart transplantation
* Instable angina pectoris/acute myocardial infarction before revascularisation
* Cardiorespiratory unstable patients
* History of valve replacement operation less than 4 weeks ago
* Obstructive cardiomyopathy with severe dynamic Left Ventricular Outflow Tract (LVOT) obstruction
* Known severe bleeding diathesis
* Known malformations or disease in the upper airways, conflicting with the catheter insertion
* Known malformations or disease in the esophagus, conflicting with the catheter insertion
* Uncontrolled arterial hypertonia (syst. blood pressure > 200mmHg)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients: Adults, hospitalised at University Hospital Bern, Dept. of Cardiology.
  Healthy subjects: Adults without any assumed or known cardiac disease.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of correct classified A/V beats in automated eECG analysis compared to manually analyzed surface ECG | during analysis of ECG (approx. 30 minutes records)

SECONDARY OUTCOMES:
Number of correctly detected atrial fibrillation sequences in automated eECG analysis compared to manually analyzed surface ECG | during analysis of ECG (approx. 30 minutes records)

CONTACTS AND LOCATIONS:
Overall Officials: Hildegard Tanner, Prof. Dr. med., Principal Investigator — Dept. of Cardiology, University Hospital Bern
Locations (1):
- Dept. of Cardiology, University Hospital Bern, Bern, Switzerland

REFERENCES:
- [Background] Haeberlin A, Niederhauser T, Marisa T, Goette J, Jacoment M, Mattle D, Roten L, Fuhrer J, Tanner H, Vogel R. The optimal lead insertion depth for esophageal ECG recordings with respect to atrial signal quality. J Electrocardiol. 2013 Mar-Apr;46(2):158-65. doi: 10.1016/j.jelectrocard.2012.12.004. Epub 2013 Jan 8. PMID 23305907
- [Background] Haeberlin A, Niederhauser T, Tanner H, Vogel R. Atrial waveform analysis using esophageal long-term electrocardiography reveals atrial ectopic activity. Clin Res Cardiol. 2012 Nov;101(11):941-2. doi: 10.1007/s00392-012-0477-6. Epub 2012 May 22. No abstract available. PMID 22614730
- [Background] Haeberlin A, Roten L, Schilling M, Scarcia F, Niederhauser T, Vogel R, Fuhrer J, Tanner H. Software-based detection of atrial fibrillation in long-term ECGs. Heart Rhythm. 2014 Jun;11(6):933-8. doi: 10.1016/j.hrthm.2014.03.014. Epub 2014 Mar 12. PMID 24632179
- [Background] Wallmann D, Tuller D, Wustmann K, Meier P, Isenegger J, Arnold M, Mattle HP, Delacretaz E. Frequent atrial premature beats predict paroxysmal atrial fibrillation in stroke patients: an opportunity for a new diagnostic strategy. Stroke. 2007 Aug;38(8):2292-4. doi: 10.1161/STROKEAHA.107.485110. Epub 2007 Jun 21. PMID 17585079
- [Derived] Wildhaber RA, Bruegger D, Zalmai N, Malmberg H, Goette J, Jacomet M, Tanner H, Haeberlin A, Loeliger HA. Estimation of the Cardiac Field in the Esophagus Using a Multipolar Esophageal Catheter. IEEE Trans Biomed Circuits Syst. 2018 Aug;12(4):791-800. doi: 10.1109/TBCAS.2018.2817027. Epub 2018 May 7. PMID 29993892